CLINICAL TRIAL: NCT03453242
Title: Age Influence on Cortical Bone Measured by Ultrasound
Acronym: OCO-US
Status: Terminated | Type: Observational
Why Stopped: Difficulty of recruitment due to COVID-19
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: K 171006J
Record Dates: First submitted 2018-01-24; First posted 2018-03-05 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Cortical Bone Erosion
Keywords: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Bone measurement by HR-pQCT and ultrasound — Measurement will be performed at radius and at tibia (ultra-distal and distal). For all the sites one measurement will be performed by HR-pQCT to get reference values of thickness and BMDs. For the distal positions and additional measurement will be performed by an innovative ultrasound device that estimates cortical thickness and porosity.

SUMMARY:
The study of this study is to evaluate the age influence on cortical bone strength properties by two methods:HR-pQCT (HighResolution-peripheral quantitativeComputedTomography) and ultrasound. The main objective consists in the evaluation of the age influence on cortical thickness at 1/3 distal radius measured by US.

DETAILED DESCRIPTION:
The study of this study is to evaluate the age influence on cortical bone by two methods: HR-pQCT and ultrasound.

84 patients will be measured. The cohort will be:

* 21 women less than 70
* 21 women more than 70
* 21 men less than 70
* 21 men more than 70 Measurement will be performed at radius and at tibia (ultra-distal and distal). For all the sites one measurement will be performed by HR-pQCT to get reference values of thickness and BMDs. For the distal positions and additional measurement will be performed by an innovative ultrasound device that estimates cortical thickness and porosity.

The participation to the study implies only a participation of one hour from the patient (30min for HR-pQCT measurements, 30 min for US).

The main objectives consist in :

* evaluating the age influence on cortical thickness at 1/3 distal radius measured by US
* evaluating the age influence on cortical thickness at distal tibia measured by US
* comparing porosities values measured by US to vBMD obtained by HR-pQCT
* comparing cortical thickness values measured by HR-pQCT at 1/3 distal radius position to ultra-distal radus position and to the tibia
* comparing vBMD values measured by HRpQCT at 1/3 distal radius position to ultra-distal radius position and to the tibia

ELIGIBILITY:
Inclusion Criteria:

* being 18 or older
* coming from the rheumatology consultation at Lariboisière Hospital

Exclusion Criteria:

* BMI > 28
* BMI < 15
* cortisone treatment
* recent fracture at non-dominant arm
* wound on measuring zone
* treatment interfering with bone architecture or bone density : oral of transdermic oestrogenes, bisphosphonates (Alendronate, Risedronate, Zoledronate) or Denosumab during the past 6 months-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort will be:
  Women and men less than 70 Women and men more than 70
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
Cortical parameters measurement | Inclusion time
  Cortical thickness at distal radius 1/3

SECONDARY OUTCOMES:
Tibia parameters measurement by US | Inclusion time
  Cortical thickness distal 1/2 tibia obtained by US
  * ultra-distal and 1/3 distal cortical thicknesses obtained by HR-pQCT
  * ultra-distal and 1/3 distal vBMD obtained by HR-pQCT
Tibia parameters measurement by HR-pQCT | Inclusion time
  Cortical thickness distal 1/2 tibia obtained by HR-pQCT
  * ultra-distal and 1/3 distal cortical thicknesses obtained by HR-pQCT
  * ultra-distal and 1/3 distal vBMD obtained by HR-pQCT
Porosity measurement | Inclusion time
  Ultrasonic porosity obtained by HR-pQCT
vBMD measurement | Inclusion time
  vBMD obtained by HR-pQCT
Cortical parameters measurement | Inclusion time
  1/3 distal cortical thicknesses obtained by HR-pQCT
Thicknesses measurement | Inclusion time
  Ultra-distal thicknesses obtained by HR-pQCT
Ultra-distal vBMD measurement | Inclusion time
  Ultra-distal vBMD and third distal obtained by HR-pQCT

CONTACTS AND LOCATIONS:
Overall Officials: Cohen-Solal Martine, Martine, Principal Investigator — APHP
Locations (1):
- Cohen-Solal, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barkmann R, Kantorovich E, Singal C, Hans D, Genant HK, Heller M, Gluer CC. A new method for quantitative ultrasound measurements at multiple skeletal sites: first results of precision and fracture discrimination. J Clin Densitom. 2000 Spring;3(1):1-7. doi: 10.1385/jcd:3:1:001. PMID 10745297
- [Background] Bochud N, Vallet Q, Bala Y, Follet H, Minonzio JG, Laugier P. Genetic algorithms-based inversion of multimode guided waves for cortical bone characterization. Phys Med Biol. 2016 Oct 7;61(19):6953-6974. doi: 10.1088/0031-9155/61/19/6953. Epub 2016 Sep 12. PMID 27617648
- [Background] Zebaze RM, Ghasem-Zadeh A, Bohte A, Iuliano-Burns S, Mirams M, Price RI, Mackie EJ, Seeman E. Intracortical remodelling and porosity in the distal radius and post-mortem femurs of women: a cross-sectional study. Lancet. 2010 May 15;375(9727):1729-36. doi: 10.1016/S0140-6736(10)60320-0. PMID 20472174